CLINICAL TRIAL: NCT02135328
Title: Somali, Latino & Hmong Radio Stories About Children's Healthy Eating and Exercise: A SoLaHmo Pilot Study
Brief Title: SoLaHmo Radio Stories About Children's Healthy Eating and Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: West Side Community Health Services (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1209S19821
Record Dates: First submitted 2014-05-05; First posted 2014-05-09 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Dietary behaviors; Physical activity behaviors; Radio story, entertainment health education; Immigrants; Somali, Latino, Hmong; Families with 3-18 year old children
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radio Story (Experimental): Participants listen to a radio story about a family's' success with preventing or managing type 2 diabetes through diet and physical activity; the focus was for the entire family to implement healthful lifestyle behaviors so the children can learn as well.
  Interventions: Behavioral: Radio Story
- Audio brochure (Active Comparator): Participants received an audio version of a standard brochure about type 2 diabetes prevention and management.
  Interventions: Behavioral: Audio brochure

INTERVENTIONS:
Behavioral: Radio Story — For the purposes of this study a "Radio Story" is an audio recorded story of about a family's success story about type 2 diabetes mellitus prevention and management.
  Arms: Radio Story
Behavioral: Audio brochure — The control participants listened to an adio version of a standard brochure about prevention and management of type 2 diabetes.
  Arms: Audio brochure

SUMMARY:
The purpose of this study is to use a community based participatory action research (CBPAR) approach to 1) create "radio stories" about Somali, Latino and Hmong families' real success stories with type 2 diabetes mellitus (DM) in managing their disease through implementation of healthful lifestyle behaviors (nutrition and physical activity), and 2) test the effectiveness and acceptability of radio stories on participant intentions to engage in or improve healthful lifestyle behaviors. Participants in the Intervention condition listened to the "radio stories" and the participants in the control condition listened to an audio brochure with relevant information. We hypothesized that the intervention participants would report higher intensions to engage in various healthful lifestyle behaviors than the control participants after both participants listened to their respective health information.

DETAILED DESCRIPTION:
Given the high rate of type 2 diabetes mellitus (diabetes) in minority and immigrant communities, implementing culturally and linguistically appropriate health promotion activities that improve families' diet and physical activity behaviors is imperative. "Radio Stories" is an education entertainment strategy that has significant potential as a health promotion tool. Through a CBPAR process, we aimed to create and test the effectiveness and acceptability of "SoLaHmo Radio Stories" about changing knowledge and behaviors to prevent or manage diabetes for Somali, Latino, and Hmong families.

Methods: SoLaHmo community researchers interview 3 families (1 Somali, 1 Latino, and 1 Hmong) who have successfully implemented lifestyle changes to prevent or manage diabetes, and then create 3 "radio stories" based on the families' experiences. To test the stories, we are conducting a two-arm trial that includes intervention groups (20 people per community) that listen to the radio stories and control groups (20 people per community) that receive a brochure with similar information (N=120). Effectiveness and acceptability of the program will be tested with pre-and post questionnaires.

Anticipated Results: Higher rates of satisfaction, increased knowledge, and intention to change in participants receiving the radio stories, as compared to control group participants, will indicate radio story program effectiveness and acceptability.

ELIGIBILITY:
Inclusion Criteria for Key Family Informant Interviews:

* Family self-identifies as Somali, Latino or Hmong
* Family has at least one child between the ages of 3-18 years old
* English or Spanish or Somali or Hmong speaking
* Family identified as having a compelling story with childhood obesity or Type 2 diabetes prevention

Inclusion Criteria for Intervention and Control Group Participants:

* Self-identified member of Somali, Latino or Hmong communities
* Adult age 18 years and older
* English or Spanish or Somali or Hmong-speaking
* Parent/caregiver is involved with raising children between the ages of 3-18 years

Exclusion Criteria for Key Family Informant Interviews:

* Family does not self-identify as Somali, Latino or Hmong
* Family does not have children between the ages of 3-18 years
* Not English or Spanish or Somali or Hmong speaking
* Parent/caregiver Is not involved with raising children between the ages of 3-18 years

Exclusion criteria for Intervention and Control Group Participants:

* Participants do not self-identify as Somali, Latino or Hmong
* Participants are younger than 18 years
* Participants are not caregivers of children between the ages of 3-18 years
* Not English or Spanish or Somali or Hmong speaking

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Acceptability and effectiveness of radio stories, a health communication intervention that addresses family eating behaviors and physical activity among immigrant Somali, Latino, and Hmong families | Intentions to change behavior from baseline to follow-up. After listening to radio story or audio brochure, an average of 25 minutes.
  The baseline and follow-up survey questions to test the "radio stories" included 15 items referring to intentions to change or improve a specific diet, physical activity, and health related behavior. There were four Likert scale response categories, from 'strongly disagree' to 'strongly agree.' In addition, the follow-up survey included questions to assess participant perceptions of the radio stories relating to their emotional connection to the story, relevance with their own experience, believability, and increase awareness and concern about type 2 diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Chrisa Arcan, Ph.D., Principal Investigator — University of Minnesota; Shannon L Pergament, MPH, MSW, Principal Investigator — West Side Community Health Services/SoLaHmo Partnership for Health and Wellness